CLINICAL TRIAL: NCT03907397
Title: Challenging to Food With Escalating Thresholds for Reducing Food Allergy
Brief Title: Immune Basis and Clinical Implications of Threshold-based Phenotypes of Peanut Allergy
Acronym: CAFETERIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scott Sicherer (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Scott Sicherer, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0722; U19AI136053 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Food Allergy; Peanut Allergy
Keywords: allergy; food; peanut; threshold; immunotherapy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: 150-200 children undergoing DBPCFC to peanut to identify 72 with high threshold peanut allergy for randomization in trial.
Masking Description: Although a double-blind, placebo controlled oral food challenge test is used in screening to identify participants eligible to continue to randomization in the study, those randomized to peanut ingestion versus avoidance have participants aware and unmasked regarding the study arm to which they were randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Ingests peanut - . Depending upon reaction threshold, participants may begin with different starting amounts of store bought peanut butter measured with study-supplied kitchen measuring spoons.
  Interventions: Biological: Peanut Protein
- Avoidance (Other): Avoids peanut, standard care
  Interventions: Other: Continued peanut avoidance

INTERVENTIONS:
Biological: Peanut Protein — up to 3 level teaspoons peanut butter or equivalent (approximately 3400 mg)
  Arms: Treatment
Other: Continued peanut avoidance — Standard of care avoidance of peanut
  Arms: Avoidance

SUMMARY:
The primary objective of this study is to determine whether allowing ingestion of sub-threshold amounts of peanut in those with a high threshold (tolerate at least 143 mg peanut protein on supervised double-blind, placebo-controlled oral food challenge [DBPCFC]) will be associated with attaining even higher thresholds over time in children with high threshold peanut allergy compared to those avoiding peanut. The secondary clinical objectives include assessing the development of sustained unresponsiveness (SU, a surrogate term for tolerance without daily ingestion), effects on quality of life, and safety compared to those avoiding peanut. Additionally, this study will phenotype the allergic response to peanut based on threshold and response to exposure. Mechanistic study objectives will determine the immune and molecular basis of the high threshold endotype, identify predictors of response to exposure, and determine mechanisms and biomarkers of remission.

ELIGIBILITY:
Inclusion Criteria:

-Subject and/or parent guardian must be able to understand and provide informed consent.

Inclusion criteria for screening DBPCFC:

* Age 4-14 years
* either sex
* any race, any ethnicity
* who are enrolled while strictly avoiding peanut
* have a history of sensitization (detectable peanut IgE >0.35 kUA/L)

Inclusion criteria for randomization:

* On screening DBPCFC are able to ingest >= 143 mg peanut protein but < 5043 mg peanut protein.
* All children will have documented consent and assent as is appropriate for age.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* Serum peanut-specific IgE antibody level > 50 kUA/L
* Recent (within the past 2 years) life-threatening (grade 3) anaphylactic reaction to peanut.
* Any disorder in which epinephrine is contraindicated such as known hypertension or cardia rhythm disorders.
* History of chronic disease requiring therapy (other than asthma, atopic dermatitis, rhinitis).
* On a build-up phase of any allergen immunotherapy.
* For those with a history of asthma, the following are assessed and any of the following is an exclusion (markers of current uncontrolled or moderate to severe asthma):

  1. FEV1 value <80% predicted (only for participants age 7 years or older and are able to perform spirometry)
  2. ACT or cACT < 20
  3. >Step 3 controller therapy as defined for children 0-4, 5-11 and >=12 years of age by EPR-3 tables
  4. Use of steroid medications in the following manners:

     1. history of daily oral steroid dosing for >1 month during the past year,
     2. having 1 burst or steroid course within the past 6 months, or
     3. having >1 burst oral steroid course within the past 12 months.
  5. Asthma requiring >1 hospitalization in the past year for asthma or >1 ED visit in the past 6 months for asthma, or any prior intubation/mechanical ventilation for asthma/wheezing.
  6. When COVID related institutional restrictions on spirometry are in effect, spirometry will not be performed and peak flow will be used with 80% predicted as cut-off.
* Gastrointestinal eosinophilic disorders, esophagitis, gastroenteritis.
* Use of short-acting antihistamines (diphenhydramine, etc.) more than one time within 3 days prior to DBPCFC or skin testing.*
* Use of medium-acting antihistamines (hydroxyzine, loratadine, etc.) more than one time within 7 days of DBPCFC or skin testing.*
* Use of systemic steroid medications (IV, IM or oral) for indications other than asthma for > 3 weeks within the past 6 months
* Use of beta-blockers (oral), (ACE) inhibitors, angiotensin-receptor blockers or calcium channel blockers.
* Participation in any trials of therapeutic interventions for food allergy in the past year.
* Therapy with anti-IgE or other biologics, including within 1 year of enrollment.
* Use of investigational drugs within 52 weeks of participation.
* Allergy to all of the following: oat, rice, corn, tapioca.
* Pregnancy
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

*Any subject meeting these criteria during the visits can be rescheduled for the oral food challenge or prick skin testing.*

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sicherer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Sicherer SH, Bunyavanich S, Berin MC, Lo T, Groetch M, Schaible A, Perry SA, Wheatley LM, Fulkerson PC, Chang HL, Suarez-Farinas M, Sampson HA, Wang J. Peanut Oral Immunotherapy in Children with High-Threshold Peanut Allergy. NEJM Evid. 2025 Mar;4(3):EVIDoa2400306. doi: 10.1056/EVIDoa2400306. Epub 2025 Feb 10. PMID 39928078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From August 2019 to April 2022 at one clinical site in the US. A total of 129 participants were assessed for eligibility and 73 fulfilled criteria for randomization.
Groups:
- Peanut Protein: Ingests peanut - . Depending upon reaction threshold, participants may begin with different starting amounts of store bought peanut butter measured with study-supplied kitchen measuring spoons.
  Peanut Protein: up to 3 level teaspoons peanut butter or equivalent (approximately 3400 mg)
Period: Overall Study
Arm/Group | Peanut Protein | Avoidance
Started | 38 | 35
Completed | 30 | 29
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 5 | 4
Not completed — withdrew after Day 1 of the primary endpoint desensitization visit. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peanut Protein | Avoidance | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 6.0 [5.0 to 10.0] | 7.0 [4.0 to 11.0] | 7.0 [5.0 to 10.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 19 | 26 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 4 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 24 | 42
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Skin prick test [Median (Inter-Quartile Range); unit: mm] — A skin test reaction is considered positive if the wheal size for the antigen is at least 3 mm larger than the wheal size of the negative control (saline).
  mm | 8.0 [6.5 to 11.0] | 9.0 [7.0 to 9.5] | 9.0 [7.0 to 10.5]
Peanut IgE level [Median (Inter-Quartile Range); unit: kUA/L] | 5.5 [2.4 to 8.7] | 4.6 [2.0 to 9.1] | 5.1 [2.1 to 8.9]
Peanut IgG4 level [Median (Inter-Quartile Range); unit: mgA/L] — Population: one sample did not have enough plasma for the IgG run.
  mgA/L
    number analyzed (Participants) | 37 | 35 | 72
    (all) | 0.4 [0.1 to 1.2] | 0.4 [0.1 to 1.4] | 0.4 [0.1 to 1.3]
Ara h2 IgE level [Median (Inter-Quartile Range); unit: kUA/L] | 3.8 [1.2 to 6.9] | 2.6 [1.5 to 6.3] | 2.9 [1.3 to 6.7]
Ara h2 IgG4 level [Median (Inter-Quartile Range); unit: mgA/L] — Population: one sample did not have enough plasma for the IgG run.
  mgA/L
    number analyzed (Participants) | 37 | 35 | 72
    (all) | 0.020 [0.007 to 0.060] | 0.050 [0.007 to 0.110] | 0.030 [0.007 to 0.100]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Children That Tolerate the Full Challenge
Description: The difference between the treatment and comparison (avoidance) groups in the percentage of children who by the endpoint double-blind, placebo-controlled oral food challenge (DBPCFC) tolerate a dose at least 2 steps higher than their baseline DBPCFC or 9043 mg of peanut protein.
  Due to missing data in the primary endpoint, the protocol & SAP specified a priori that missing data would be imputed using multiple imputation and results based on 30 completed-imputed data sets would be combined using Rubin's rule. In the Peanut Protein group, the observed data was so strong that participants with missing data were also imputed as success across all imputations (hence, 100% success rate). In the Peanut Avoidance group, there was more variability in the proportion of successes across imputations and these varying proportions were averaged. Missing data were imputed and results were pooled.
Time Frame: 72 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
percentage of participants | 100 | 21

2. Secondary Outcome: The Percentage of Children That Achieve Sustained Unresponsiveness
Description: The percentage of children who achieve sustained unresponsiveness or natural tolerance during the study.
Time Frame: 96 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
percentage of participants | 68.4 [53.6 to 83.2] | 8.6 [0 to 17.9]

3. Secondary Outcome: Number of Children With Acute Allergic Reactions
Description: Safety parameter assessed by number of participants with acute allergic reactions which includes anaphylaxis or gastrointestinal side effects.
Time Frame: 96 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
Participants | 25 | 11

4. Secondary Outcome: Mean Change in Food Allergy Quality of Life Parental Burden Instrument
Description: The Food Allergy Quality of Life-Parental Burden (FAQL-PB) Scale is a 17-item instrument. It utilizes a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). The number circled for each question is summed to provide a total continuous score range of 0 to 102 with a higher score indicating greater burden on the family.
Time Frame: baseline and at 72 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
score on a scale | -7.78 [-13.10 to -2.47] | -9.23 [-14.71 to -3.74]

5. Secondary Outcome: Mean Change in SPT Wheal Size
Description: Change in Skin Prick Test (SPT) mean wheal size at 72 weeks as compared to baseline. A skin test reaction is considered positive if the wheal size for the antigen is at least 3 mm larger than the wheal size of the negative control (saline).
Time Frame: Baseline and 72 weeks
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
mm | -3.05 [-4.27 to -1.84] | -0.48 [-1.74 to 0.78]

6. Secondary Outcome: Mean Change in Peanut-specific IgE
Description: Mean Change in Peanut-specific IgE level at week 72 as compared to baseline.
Time Frame: Baseline and 72 weeks
Measure: Mean (95% Confidence Interval); unit: kUA/L
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
kUA/L | -0.22 [-0.45 to 0.02] | 0.40 [0.15 to 0.64]

7. Secondary Outcome: Mean Change in Peanut-specific IgG4
Description: Mean Change in Peanut-specific IgG4 level at week 72 as compared to baseline.
Time Frame: Baseline and 72 weeks
Measure: Mean (95% Confidence Interval); unit: mgA/L
Arm/Group | Peanut Protein | Avoidance
Number analyzed (Participants) | 38 | 35
mgA/L | 3.11 [2.41 to 3.81] | 0.52 [-0.20 to 1.24]

ADVERSE EVENTS:
Time Frame: 96 weeks
Arm/Group | Peanut Protein | Avoidance
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 25/38 | 11/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peanut Protein (N=38) | Avoidance (N=35)
Abdominal Discomfort (Gastrointestinal disorders) | 9 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oral Pruritus (Gastrointestinal disorders) | 17 | 8
Vomiting (Gastrointestinal disorders) | 8 | 2
Vomiting Projectile (Gastrointestinal disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 2
Lip Edema (Immune system disorders) | 1 | 1
Pruritus Allergic (Immune system disorders) | 1 | 4
Urticaria (Immune system disorders) | 10 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Throat Tightness (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT03907397/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT03907397/SAP_001.pdf
  • Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03907397/ICF_002.pdf